CLINICAL TRIAL: NCT05218109
Title: Non-pharmacological Interventions to Improve Stress and Sleep Among College Students
Brief Title: Stress and Sleep Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB202101724
Record Dates: First submitted 2022-01-03; First posted 2022-02-01 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Stress, Psychological; Sleep; Transcutaneous Electric Nerve Stimulation; Vagus Nerve Stimulation; Mindfulness
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- tVNS + mindfulness (Experimental): Transcutaneous vagus nerve stimulation plus behavioral: mindfulness
  Interventions: Device: tVNS; Behavioral: Mindfulness
- Sham + mindfulness (Sham Comparator): Sham transcutaneous vagus nerve stimulation plus behavioral: mindfulness
  Interventions: Behavioral: Mindfulness; Device: sham tVNS
- Mindfulness only (Active Comparator)
  Interventions: Behavioral: Mindfulness
- Control (Active Comparator): Control number puzzle task delivered via mobile device
  Interventions: Other: Number Puzzle

INTERVENTIONS:
Device: tVNS — transcutaneous vagus nerve stimulation
  Arms: tVNS + mindfulness
Behavioral: Mindfulness — Brightmind mobile mindfulness application
  Arms: Mindfulness only; Sham + mindfulness; tVNS + mindfulness
Device: sham tVNS — sham transcutaneous vagus nerve stimulation
  Arms: Sham + mindfulness
Other: Number Puzzle — Control number puzzle task delivered via mobile device
  Arms: Control

SUMMARY:
This between-subject, longitudinal pilot study in healthy college students aims to explore the acceptability and preliminary outcomes of two novel and complementary interventions that may improve stress and sleep: transcutaneous vagus nerve stimulation (tVNS) and a mobile mindfulness intervention.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student (ages 18-30)
* Must own a smartphone
* Must be able to read and write English

Exclusion Criteria:

* Major medical illnesses including diagnosed severe neurological illnesses (e.g., stroke, seizure history), medical conditions associated with neurological effects (e.g. heart, kidney disease), autoimmune disorders, and severe psychiatric diseases (e.g., schizophrenia)
* Pregnancy
* History of brain surgery, tumor, intracranial metal implantation, pacemakers or other implanted devices
* History of adverse reaction to electrical nerve stimulation
* Prescribed sleep medications and/or psychotropic medications
* Illicit or prescription drug abuse within the last two months (marijuana or alcohol abuse >2 weeks out will be acceptable for inclusion)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bottari, M.S., Principal Investigator — University of Florida; Liva LaMontagne, Dr. Psych., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to study arms/groups pseudo-randomly upon scheduling an intake appointment (prior to enrollment).
Period: Overall Study
Arm/Group | tVNS + Mindfulness | Sham + Mindfulness | Mindfulness Only | Control
Started | 16 | 20 | 20 | 20
Week 1 | 14 | 15 | 19 | 20
Week 2 | 13 | 14 | 19 | 20
Week 3 | 12 | 13 | 19 | 18
Week 4 | 13 | 14 | 19 | 19
Week 8 (Follow Up) | 14 | 14 | 17 | 20
Completed | 14 | 14 | 17 | 20
Not Completed | 2 | 6 | 3 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant in the tVNS + mindfulness group and 3 participants in the sham + mindfulness group were screened out of the study during the intake visit after enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | tVNS + Mindfulness | Sham + Mindfulness | Mindfulness Only | Control | Total
Number analyzed (Participants) | 15 | 17 | 20 | 20 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.67 (2.38) | 19.71 (1.26) | 19.95 (1.73) | 20.75 (1.45) | 20.26 (1.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 10 | 10 | 42
  Male | 5 | 5 | 10 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 8 | 9 | 23
  Not Hispanic or Latino | 11 | 15 | 12 | 11 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 7 | 5 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2 | 4
  White | 9 | 6 | 9 | 10 | 34
  More than one race | 1 | 1 | 2 | 1 | 5
  Unknown or Not Reported | 2 | 2 | 3 | 4 | 11
Pittsburg Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: units on a scale] — The PSQI (Buysse et al., 1989) contains 19 self-rated items that are combined to form seven component scores, each of which has a range from 0-3 points. For each component, a score of 0 indicates no difficulty, while a score of 3 indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range from 0-21 points (0 = best sleep quality, 21 = poorest sleep quality).
  units on a scale | 8.13 (2.70) | 9.29 (2.71) | 8.9 (2.61) | 7.25 (3.00) | 8.38 (2.83)
Perceived Stress Scale (PSS) [Mean (Standard Deviation); unit: units on a scale] — The PSS (Cohen et al., 1994) is a 10-item questionnaire measuring the degree to which situations in one's life are appraised as stressful. In particular, it gauges how unpredictable, uncontrollable, and overloaded respondents find their lives. Participants rate each item on a scale of 0 (never) to 4 (very often), and total scores range from 0-40 (0 = least perceived stress, 40 = most perceived stress).
  units on a scale | 14.87 (5.59) | 16.47 (7.26) | 14.80 (5.15) | 16.35 (6.00) | 15.64 (5.95)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Combined tVNS + Mindfulness Intervention as Assessed by Participant Self-report of Acceptability Using the Acceptability of Intervention Measure (AIM)
Description: The AIM (Weiner et al., 2017) is a brief 4-item scale measuring the degree to which participants believe an intervention is acceptable. The response scale for each item ranges from 1 (completely disagree) to 5 (completely agree). Responses from the 4 items are averaged to yield total scores ranging from 1-5, with higher scores indicating greater acceptability.
Time Frame: Assessed in the tVNS + mindfulness groups and sham + mindfulness groups at Week 2
Population: Enrolled participants in the tVNS + mindfulness groups and sham + mindfulness groups who completed the Week 2 questionnaires at the appropriate timeframe were included in the analysis. Results are not reported for the Mindfulness only and Control groups, as these participants did not receive the tVNS portion of the combined intervention. Therefore, they did not complete the AIM measure asking about acceptability of the tVNS intervention and data was not available to report on for those groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tVNS + Mindfulness | Sham + Mindfulness
Number analyzed (Participants) | 12 | 14
units on a scale | 4.08 (0.40) | 3.37 (1.15)

2. Primary Outcome: Sleep Quality as Assessed by Participant Self-report on the Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI (Buysse et al., 1989) contains 19 self-rated items that are combined to form seven component scores, each of which has a range from 0-3 points. For each component, a score of 0 indicates no difficulty, while a score of 3 indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range from 0-21 points (0 = best sleep quality, 21 = poorest sleep quality).
Time Frame: Assessed at the end of the intervention phase (Week 4)
Population: Enrolled participants who completed the Week 4 questionnaires during an appropriate timeframe were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tVNS + Mindfulness | Sham + Mindfulness | Mindfulness Only | Control
Number analyzed (Participants) | 13 | 14 | 19 | 19
units on a scale | 6.23 (2.62) | 8.29 (2.61) | 7.84 (2.32) | 8.21 (2.78)

3. Primary Outcome: Perceived Stress as Assessed by Participant Self-report on the Perceived Stress Scale (PSS)
Description: The PSS (Cohen et al., 1994) is a 10-item questionnaire measuring the degree to which situations in one's life are appraised as stressful. In particular, it gauges how unpredictable, uncontrollable, and overloaded respondents find their lives. Participants rate each item on a scale of 0 (never) to 4 (very often), and total scores range from 0-40 (0 = least perceived stress, 40 = most perceived stress).
Time Frame: Assessed at the end of the intervention phase (Week 4)
Population: Enrolled participants who completed the Week 4 questionnaires during the appropriate timeframe were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tVNS + Mindfulness | Sham + Mindfulness | Mindfulness Only | Control
Number analyzed (Participants) | 13 | 14 | 19 | 19
units on a scale | 11.46 (5.81) | 13.36 (6.34) | 14.47 (5.58) | 16.42 (8.66)

ADVERSE EVENTS:
Time Frame: During participants' active participation in the study (4 weeks)
Arm/Group | tVNS + Mindfulness | Sham + Mindfulness | Mindfulness Only | Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/16 | 3/20 | 0/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tVNS + Mindfulness (N=16) | Sham + Mindfulness (N=20) | Mindfulness Only (N=20) | Control (N=20)
Uncomfortable variation in stimulation intensity at stimulation site (Product Issues) | 0 (0) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT05218109/Prot_SAP_001.pdf